CLINICAL TRIAL: NCT03656952
Title: A PHASE 1, RANDOMIZED, PLACEBO-AND POSITIVE-CONTROLLED CROSSOVER STUDY TO DETERMINE THE EFFECT OF SINGLE-DOSE PF-06700841 ON QTC INTERVAL IN HEALTHY VOLUNTEERS
Brief Title: A Study to Evaluate the PF-06700841 Effect on QTc Interval in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B7931019; 2018-001932-23 (EudraCT Number)
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: PF-06700841; QT effect; concentration-QTc analysis
MeSH Terms: interventions — PF-06700841; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Seq 1 (Experimental): PF-06700841-> placebo-> moxifloxacin
  Interventions: Drug: PF-06700841; Drug: Placebo; Drug: moxifloxacin
- Seq 2 (Experimental): PF-06700841->moxifloxacin->placebo
  Interventions: Drug: PF-06700841; Drug: Placebo; Drug: moxifloxacin
- Seq 3 (Experimental): Placebo->PF-06700841->moxifloxacin
  Interventions: Drug: PF-06700841; Drug: Placebo; Drug: moxifloxacin
- Seq 4 (Experimental): Placebo->moxifloxacin->PF-06700841
  Interventions: Drug: PF-06700841; Drug: Placebo; Drug: moxifloxacin
- Seq 5 (Experimental): Moxifloxacin->PF-06700841->placebo
  Interventions: Drug: PF-06700841; Drug: Placebo; Drug: moxifloxacin
- Seq 6 (Experimental): Moxifloxacin->placebo->PF-06700841
  Interventions: Drug: PF-06700841; Drug: Placebo; Drug: moxifloxacin

INTERVENTIONS:
Drug: PF-06700841 — a single oral dose of 200 mg PF-06700841
Drug: Placebo — Placebo matching PF-06700841
Drug: moxifloxacin — a single oral dose of 400 mg moxifloxacin

SUMMARY:
A phase 1, 6-sequence, 3-period, subject- and investigator blinded and sponsor-open, crossover study in healthy volunteers to evaluate the PF-06700841 effect on QTc interval. Each subject randomized will receive placebo, PF-06700841 200 mg and moxifloxacin (open label) in one of the 6 sequences. Moxifloxacin is positive control to demonstrate the study sensitivity and PF-06700841 effect on QTc will be assessed by concentration-QT analysis

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential and/or male subjects. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including BP and pulse rate measurement, 12-lead ECG, or clinical laboratory tests.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb) at screening.
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic (including alcoholic liver disease, nonalcoholic steatohepatitis (NASH), autoimmune hepatitis, and hereditary liver diseases), psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing)
* Self-reported history or risk factors for QT prolongation or torsades de pointes (eg, organic heart disease, congestive heart failure, hypokalemia, hypomagnesaemia, congenital long QT syndrome, myocardial ischemia or infarction), congenital deafness, family history of sudden death, and family history of long QT syndrome.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product (whichever is longer)
* Subjects with known prior participation (ie, randomized and received at least 1 dose of investigational product) in a trial involving PF-06700841
* History of tuberculosis or active or latent or inadequately treated infection, positive QuantiFERON- tuberculosis (TB) Gold test
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb)
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
QTc change from baseline following PF-06700841 treatment | 0 to 48 hours post-dose
  QTc change from baseline at geometric mean of maximum concentrations observed after single doses of 200 mg PF-06700841 and maximum concentrations expected at lower doses of 30 and 60 mg.

SECONDARY OUTCOMES:
QTc change from baseline following moxifloxacin treatment | 0-48 hours post-dose
  QTc change from baseline at 3 hours (Tmax) after a single dose of 400 mg moxifloxacin administration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Hughes JH, Qiu R, Banfield C, Dowty ME, Nicholas T. Population Pharmacokinetics of Oral Brepocitinib in Healthy Volunteers and Patients. Clin Pharmacol Drug Dev. 2022 Dec;11(12):1447-1456. doi: 10.1002/cpdd.1163. Epub 2022 Aug 31. PMID 36045513
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7931019&StudyName=A+Phase+1%2C+Randomized%2C+Placebo+And+Positive+Controlled+Crossover+Study+To+Determine+The+Effect+Of+Single+Dose+Pf+06700841+On+Qtc+Interval+In+Healthy+Volunteers
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7931019&StudyName=A+Phase+1%2C+Randomized%2C+Placebo-and+Positive-controlled+Crossover+Study+To+Determine+The+Effect+Of+Single-dose+Pf-06700841+On+Qtc+Interval+In+Healthy+Volunteers